CLINICAL TRIAL: NCT03641729
Title: Feasibility and Safety of a Novel Individualized In-hospital Exercise Training Program for Patients Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Physical Exercise for Hematopoietic Stem Cell Transplantation (HSCT)
Acronym: HSCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Juiz de Fora (Other)
Responsible Party: Principal Investigator, Aline Priori Fioritto, Principal Investigator/ Post-Graduation Program on Collective Health, Federal University of Juiz de Fora
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2,030,132
Record Dates: First submitted 2018-08-14; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Physical Activity
Keywords: hematopoietic stem cell transplantation; exercise training; feasibility; safety
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The exercise training program was performed once daily during the hospital stay. The program included 2- to 5-minute warm-up session which consisted of stretching, coordination and balance exercises, followed by 10 to 20 minutes of moderate-intensity aerobic exercise using a lower limb cycle ergometer (Live up Sports, 1023, Araucária, Paraná, LS9055). Participants also performed three sets of five to ten repetitions of sit-to-stand exercises with a 1-minute rest interval between each set. A cool-down period of 2- to 5-minutes of stretching and breathing exercises was delivered at the end of the exercise session. All exercises were performed within the participant's room. The aerobic training target zone was set at 50% to 70% of heart rate (HR) reserve. The HR reserve was estimated using the following equation: [(220-age in years) - resting HR] x [50 to 70%] + resting HR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Patients were eligible if they were aged 18 years or older, referred for HSCT and admitted to the Bone Marrow Transplant Unit (BMTU). Patients were screened in the BMTU admission and recruited to the study after avaliation in the first-day internation.
  Interventions: Other: individualized exercise training program

INTERVENTIONS:
Other: individualized exercise training program — The exercise training program was performed once daily, included 2- to 5-minute warm-up session (stretching, coordination and balance exercises), 10 to 20 minutes of moderate-intensity aerobic exercise using a cycle ergometer, 3 - to 5-sets to ten repetitions of sit-to-stand exercises with a 1-minute rest interval between each set. A cool-down period of 2- to 5-minutes of stretching and breathing exercises was delivered at the end of the exercise session. The aerobic training target zone was set at 50% to 70% of heart rate (HR) reserve.

SUMMARY:
Objective: To evaluate whether a novel individualized exercise training program for hospitalized patients undergoing hematopoietic stem cell transplantation (HSCT) is feasible and safe and whether it would improve functional capacity, muscle strength and health-related quality of life (HRQoL).

Design: Prospective, within-group, feasibility intervention study. Setting: Bone marrow transplant unit in a general hospital. Subjects: Patients electively hospitalized for HSCT who were admitted to the bone marrow transplant unit.

Intervention: Participants performed the individualized in-hospital exercise training program on a daily basis during their hospital admission. The exercise training program was performed once a day for 20 to 40 minutes and included a warm-up period, moderate-intensity aerobic exercise (10 to 20 minutes ), muscle strengthening exercise and cool-down activities.

Outcome measures: The primary outcomes were feasibility (consent rate, attrition rate and exercise adherence) and the safety of the exercise program. Secondary outcomes included functional capacity (step test), peripheral muscle strength (sit-to-stand test) and HRQoL (QLQ-C30) were evaluated at baseline (on admission to hospital) and prior to hospital discharge.

DETAILED DESCRIPTION:
This was a prospective, within-group, feasibility intervention study which took place at the Juiz de Fora University Hospital (HU-JF) between June 2016 and June 2017.

Patients were screened in the Bone Marrow Transplant Unit (BMTU) admission and recruited to the study after avaliation in the first-day internation. However, included at study or no, all patients that had the indication (at any time during internation) received the intervention. This study was approved by the Institutional Ethics Committee (protocol: 2,030,132). All participants provided written informed consent prior to participation.

The exercise training program was performed once daily during the hospital stay. The program included 2- to 5-minute warm-up session which consisted of stretching, coordination and balance exercises, followed by 10 to 20 minutes of moderate-intensity aerobic exercise using a lower limb cycle ergometer (Live up Sports, 1023, Araucária, Paraná, LS9055). Participants also performed three sets of five to ten repetitions of sit-to-stand exercises with a 1-minute rest interval between each set. A cool-down period of 2- to 5-minutes of stretching and breathing exercises was delivered at the end of the exercise session. All exercises were performed within the participant's room. The aerobic training target zone was set at 50% to 70% of heart rate (HR) reserve. The HR reserve was estimated using the following equation: [(220-age in years) - resting HR] x [50 to 70%] + resting HR.

The indication, contraindication or interruption criteria of the exercise training program were evaluated daily based on the participant's clinical, hemodynamic and hematological parameters as described in Table 1. These parameters were recorded at rest and monitored during the intervention. The daily clinical assessment for exercise performance is described in the flowchart shown in Figure 1. A platelet count of < 10,000 cells/mm3 (cells per cubic millimeter), hemoglobin (Hb) < 7 g/dL (grams per deciliter) and/or hematocrit (Ht) < 20% were considered contraindications for the exercise program. If participants were clinically stable, they were encouraged to perform breathing exercises in bed; maintain Basic Activity of Daily Living (BADLs), which consist mostly of self-care tasks including showering, dressing and feeding; perform the individualized in-hospital exercise training program, including a moderate intensity aerobic training without or with cycle ergometer load, based on platelets, hematocrit and hemoglobin count.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for this study if they were aged 18 years or older
* And referred for HSCT and admitted to the Bone Marrow Transplant Unit (BMTU).

Exclusion Criteria:

* Patients were excluded if they were re-admitted to the hospital due to post-HSCT complications (infection, respiratory/cardiovascular complications, graft-versus-host disease - GVHD)
* Or diagnosed with any orthopedic and/or cognitive limitations that constrained the study assessments and/or training participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
recruitment rates | up to 4 weeks
  recruitment rates was considered as the acceptance rate of patients eligible for the intervention to participate in the exercise regime - goal 60%
attrition rates | up to 4 weeks
  attrition rates was considered as the acceptance rate of patients eligible for the intervention to participate in the exercise regime - until 30%
exercise adherence rates | up to 4 weeks
  exercise adherence rates was assessed as the total number of minutes the participants performed the aerobic exercise in relation to the planned exercise time of at least 70%.
adverse events rates | up to 4 weeks
  Safety of the intervention was considered if the adverse events rates was less than 5%

SECONDARY OUTCOMES:
Functional capacity | up to 4 weeks
  evaluated using the 6-minute step test (6ST)
Lower limb muscle strength | up to 4 weeks
  Lower limb muscle strength was assessed using the sit-to-stand test (STS)
Upper limb muscle strength | up to 4 weeks
  Upper limb muscle strength was assessed using a handgrip dynamometer (Sammons Preston Rolyan, 4 Sammons Court, Bolingbrook, IL 60440)
Health-related quality of life (HRQoL) | up to 4 weeks
  The European Organization for Research and Treatment of Cancer's Quality of Life Questionnaire (EORTC QLQ-C30) was used to evaluate HRQoL. The questionnaire has three domains, including overall health, functional health and symptoms, with scores ranging from 0 to 100. Higher scores in the overall and functional health domains correspond to better quality of life, while higher scores on the symptoms scale correspond to worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: FIORITTO, Principal Investigator — Federal University of Juiz de Fora

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: More information contact the principal investigator — http://aline.priori.fioritto@gmail.com
- Available data/document: Study Protocol — http://aline.priori.fioritto@gmail.com — More information contact the principal investigator